CLINICAL TRIAL: NCT04159987
Title: A Multicenter, Interventional, Open-label Study to Monitor the Evolution of Motor Function in SMA Type II Adults Patients Treated With SPINRAZA®
Brief Title: Monitoring to the Evolution of Motor Function in SMA Type II Adults Patients Treated With SPINRAZA®
Acronym: SMAII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-PP-09
Record Dates: First submitted 2019-10-04; First posted 2019-11-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal muscular atrophy patient (Experimental)
  Interventions: Other: Spinraza intrathecal injection

INTERVENTIONS:
Other: Spinraza intrathecal injection — The aim is to monitor the evolution of the Motor Function Measure-32 for SMA type II adult patients treated with SPINRAZA® (Nusinersen).

SUMMARY:
SPINRAZA® (Nusinersen) is the first intrathecal administered drug which was approved by the FDA to treat SMA children and adults (2016). The aim is to monitor the evolution of the Motor Function Measure-32 for SMA type II adult patients treated with SPINRAZA® (Nusinersen).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with SMA type II disease who are wheelchair bound,
* Must be 18 years or older,
* Men or Women with SMA type II disease (age at symptoms onset: >6 months old and who never acquired the capacity to walk but acquired the ability to sit without support) with genetic confirmed diagnosis of 5q SMA homozygous gene deletion (SMN1 exon 7/8) or mutation or compound heterozygous mutation - performed by PCR amplification and restriction digest of DNA using primers flanking SMN1 and SMN2 exon 7.
* MFM 32 score ≥ 19/96
* Lumbar CT scan showing the feasibility of intrathecal injection.
* Written informed consent from the subject prior to initiation of any study-mandated procedures
* Females of childbearing potential must have a negative pregnancy test at Screening and at Enrollment, must agree to use reliable method of contraception (if sexually active) from screening up to study drug discontinuation plus 180 days.

Exclusion Criteria:

* Patients with a high risk for thrombocytopenia or hemorrhage or renal diseases: Urine protein, platelet count and coagulation tests will be done prior to intrathecal injection with SPINRAZA®
* Patients with high risk of hydrocephalus
* Adult patients under guardianship
* Pregnant and/or breastfeeding females
* Subject has received any investigational therapy or pharmacological treatment for SMA one month prior the beginning of the study
* Subject has received gene therapy for SMA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the Motor Function Measure-32 (MFM-32) from Baseline (M0) to 1 month (M1), 3 months (M3), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  Within MFM-32, 32 terms will be evaluated to describe patient's motor functions and grouped into 3 sub-scores at baseline (M0), M1, M3, M7, M15 and M27:
  * D1: standing position and transfer
  * D2: axial and proximal motor function
  * D3: distal motor function The MFM-32 ratings rely on the use of a 4-point Likert scale based on the subject's maximal abilities without assistance (0: cannot initiate the task or maintain the starting position; 1: performs the task partially; 2: performs the task incompletely or imperfectly; 3: performs the task fully and normally.)

SECONDARY OUTCOMES:
Change of the pulmonary function, specially Force Vital Capacity (FVC%), from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  Force Vital Capacity (FVC%)will be measured in sitting position and optionally in lying position.
Change of the pulmonary function, specially Maximal Inspiratory Pressure (MIP) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  Maximal Inspiratory Pressure (MIP) will be measued in sitting position and optionally in lying position.
Change of the pulmonary function, specially Maximum Expiratory Pressure (MEP) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  Maximum Expiratory Pressure (MEP) will be measured in sitting position and optionally in lying position.
Change of the Fatigue Severity Scale (FSS) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  The FSS is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree".
Change of the Pinch and Grip test from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  The purpose of those tests is to measure the maximum isometric strength of the hand and forearm muscles when doing a grasping or a pinching action. The equipment required for the grip and the pinch tests is a calibrate dynamometer. The subject should be strongly encouraged to give a maximum effort. We record three trials for each hand, alternating hands with at least 30 seconds recovery between each effort. We keep the best result.
Change of the Repeated nine-hole peg test (r9HPT) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  The r9HPT is a modification of the 9-Hole Peg test (9HPT) targeting endurance instead of motor function. The 9HPT is a brief, standardized, quantitative test of upper extremity function.
  In r9HPT, participants performed 5 consecutive rounds of the 9HPT, without break, using the same and preferred hand. We will look at the change (ratio) in score between the last trial and the first trial, an increase in time needed to perform the test in consecutive rounds indicating the apparition of the muscle fatigability.
Change of the Revised Hammersmith Scale (RHS) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  The RHS consisted of 36 items for very weak SMA 2 through to very strong SMA 3. With regards scoring, 33 items were graded on an ordinal scale of 0, 1, 2 (where 0 denotes the least level of ability/function progressing to the highest level of ability to achieve a score of 2), the remaining 3 items were scored 0, 1 (where 0 is unable and 1 was able to achieve). The maximum achievable score is 69.
Change of the Iowa Oral Performance Instrument (IOPI) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27 | at baseline, 1, 3, 7, 15 and 27 months
  The Iowa Oral Performance Instrument (IOPI) is a means to quantify lip, tongue, and buccal strength using a validated tool with published ranges for normative data for lingual measurements
Change of the Revised Upper Limb Module (RULM) from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27 | at baseline, 1, 3, 7, 15 and 27 months
  The RULM is a validated measure and used only for patients with SMA that evaluates shoulder, wrist, and hand functions. It takes approximately 15 minutes to administer and requires a toolkit that is used to have the patient repeat specific tasks (eg, picking up a coin, bringing hand to mouth) with both arms. RULM is a scale of 19 scorable items; each item is scored from 0 to 2:
  * 0=Unable
  * 1=Able, with modification
  * 2=Able, no difficulty The maximum score is 37 and the patients are scored on both upper limbs.
Change of the Electrophysiological assessment, specially Motor Unit Number Index (MUNIX), from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  MUNIX is a neurophysiologic test which provide an index of functioning lower motor neurons in a muscle. MUNIX total score is calculated by adding the individual values of the 6 tested muscles (abductor pollicis brevis, abductor digiti minimi, first dorsal interosseous, deltoid, tibialis anterior and trapezius).
Change of the Electrophysiological assessment, specially Motor Units Size Index (MUSIX), from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27) | at baseline, 1, 3, 7, 15 and 27 months
  MUSIX is a neurophysiologic tests which provide an index of functioning lower motor neurons in a muscle. MUSIX is calculated by dividing MUNIX by the Compound Motor Action Potential (CMAP) amplitude, measured in 6 tested muscles (abductor pollicis brevis, abductor digiti minimi, first dorsal interosseous, deltoid, tibialis anterior and trapezius).
Change of the health Status from Baseline (M0) to 1 month (M1), 7 months (M7), 15 months (M15) and 27 months (M27 | at baseline, 1, 3, 7, 15 and 27 months
  Health Status will be assessed using the question quality of Life in genetic Neuromuscular Disease (QoL-gNMD), specifically designed for patients with a slowly-progressive neuromuscular disease with genetic predominant muscular damage. The QoL-gNMD is splitted in 3 domains: "Impact of Physical Symptoms" (score from 0 to 19), "Self-perception" (score from 0 to 24) and "Activities and Social Participation" (score from 0 to 27).

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU de Lyon, Lyon, Auvergne-Rhône-Alpes
  - CHRU de Lille, Lille, Hauts-de-France
  - CHU de Montpellier, Montpellier, Occitanie
  - CHU de Toulouse, Toulouse, Occitanie
  - Hopital de la Timone - APHM, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region
  - APHP, Paris, Île-de-France Region